CLINICAL TRIAL: NCT01271075
Title: Double-blind, Triple Cross-over, Placebo-controlled Study to Assess the Efficacy, Mechanisms, and Safety of Treatment With Bilastine 20 mg, 40 mg and 80 mg in Cold Contact Urticaria (CCU)
Brief Title: Bilastine Updosing - Characterization of Underlying Mechanisms
Acronym: BUCUM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Faes Farma, S.A. (Industry)
Responsible Party: Principal Investigator, Karoline Krause, Karoline Krause, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BUCUM 2010; 2010-019344-39 (EudraCT Number)
Record Dates: First submitted 2010-12-30; First posted 2011-01-06 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Cold Contact Urticaria
Keywords: urticaria; bilastine
MeSH Terms: conditions — Cold Urticaria; Urticaria | interventions — bilastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilastine A (Active Comparator): A: Crossover Bilastine 20 mg, Bilastine 40 mg, Placebo, Bilastine 80 mg
  Interventions: Drug: Bilastine
- Bilastine B (Active Comparator): B: Crossover Bilastine 80 mg, Placebo, Bilastine 40 mg, Bilastine 20 mg
  Interventions: Drug: Bilastine

INTERVENTIONS:
Drug: Bilastine — Single dose, oral, 20 mg, 40 mg, 80 mg each for 7 days
  Arms: Bilastine A
Drug: Bilastine — Single dose, oral, 20 mg, 40 mg, 80 mg each for 7 days
  Arms: Bilastine B

SUMMARY:
This is a double-blind, triple cross-over, placebo-controlled study to assess the efficacy, mechanisms, and safety of treatment with the antihistamine bilastine in patients with cold contact urticaria (CCU).

Efficacy is primarily assessed by a change in critical stimulation time thresholds (CSTT) and critical temperature thresholds (CTT) after treatment with different dosages of bilastine (20 mg, 40 mg, 80 mg). Following a baseline period of 2-4 weeks, patients are randomized to either group A or group B. In group A they are given bilastine 20 mg, 40 mg, placebo and bilastine 80 mg for 7 days each followed by a 14-day washout period at a time. In group B they are given bilastine 80 mg, placebo, 40 mg and 20 mg for 7 days each followed by a 14-day washout period at a time. CSTT and CTT testings are performed at each of 6 visits, skin microdialysis for the assessment of mast cell mediators is performed at V2, V3 and V6. Visits for investigator's assessments are scheduled at day -14 to -28, day 0, day 7, day 28, day 49, and day 70. Overall a max. of 20 subjects with cold contact urticaria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Reliable method of contraception for both women of childbearing potential as well as man during the study and 3 months thereafter. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner
* Outpatients with CCU for more than 6 weeks. Urticaria symptoms must comprise wheal and itch.
* Age above 18 years.
* No participation in other clinical trials 1 months before and after participation in this study

Exclusion Criteria:

* Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1, number 4 AMG (Arzneimittelgesetz)
* The presence of permanent severe diseases, especially those affecting the immune system, except urticaria and cold urticaria
* The presence of permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
* History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
* ECG alterations of repolarisation (QTc prolongations > 450ms)
* Blood pressure >180/100 mmHg and/or heart rate >100/min.
* Evidence of significant hepatic or renal disease (GOT and/or GPT 3 times above the upper reference value, serum creatinine 1.5 times above the upper reference value)
* History of adverse reactions to bilastine or known hypersensitivity to bilastine or its ingredients
* Presence of active cancer which requires chemotherapy or radiation therapy
* Presence of alcohol abuse or drug addiction
* Intake of oral corticosteroids within 14 days prior to screening visit
* Use of depot corticosteroids or chronic systemic corticosteroids within 21 days prior to screening visit
* Use of systemic immunosupressants/immunomodulators like ciclosporine A, dapsone, methotrexate, mycophenolate, chloroquine, and comparable drugs within 28 days prior to screening visit
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The effects of a standard dose (20 mg) and higher than standard doses of bilastine (40 mg and 80 mg) on symptom development in CCU patients | 6 visits in 12-14 weeks
  Change in critical stimulation time thresholds (CSTT) and critical temperature thresholds (CTT) after treatment with different dosages of bilastine (20 mg, 40 mg, 80 mg).

SECONDARY OUTCOMES:
The effects of a standard dose (20 mg) and higher than standard doses of bilastine (80 mg) on mast cell mediator release in CCU patients | Visit 2 (day 0), visit 3 (day 7) and visit 6 (day 70)
  Change in mast cell mediator release, including histamine and mast cell-derived cytokines (e.g. IL-1, IL-6, IL-8, IL-13, TNF) after standard dose treatment with bilastine (20 mg) compared to high dose bilastine (80 mg) and baseline.
Safety and tolerability following administration of bilastine to patients with cold contact urticaria | up to 14 weeks
  Safety and tolerability: This includes physical examination, routine safety laboratory assessments, clinical observation, vital signs and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany